CLINICAL TRIAL: NCT06126185
Title: Synbiotic Treatment for Neuropsychiatric Symptom of Autism Spectrum Disorder: an Open-label Pilot Study
Brief Title: Open-label Pilot Study Synbiotic Treatment for Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Wing Ho, Assistant Professor (Clinical), Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023.484
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder; Anxiety
Keywords: synbiotic; probiotic; prebiotic
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Synbiotic treatment (Experimental): 12-week course of synbiotic
  Interventions: Dietary Supplement: 12-week course of synbiotic

INTERVENTIONS:
Dietary Supplement: 12-week course of synbiotic — A 12-week-course of synbiotic, which contains containing 5 billion colony-forming unit (CFU) of a combination of 4 probiotic species belonging to the genus of Lactobacillus, Bifidobacterium and Streptococcus, and 3 prebiotics, will be given to participants to take daily through oral route.

SUMMARY:
The objective of this study is to conduct a open-label pilot study evaluating the feasibility, tolerability and preliminary efficacy of a 12-week course of synbiotic in improving anxiety symptoms in children with ASD. The investigators hypothesise that the course of synbiotic will feasible and tolerable, and that there will be a reduction in anxiety symptoms in ASD children after the 12-week course of synbiotic.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a neurodevelopmental disorder defined by the core features of social communication deficits and restricted and repetitive behaviour (RRB). One important treatment target of ASD children is co-occurring neuropsychiatric disorders, which would interact with the core symptoms to further jeopardize their social and educational development. In pre-pubertal children, anxiety disorder is one of the commonest co-occurring psychiatric disorders without effective therapeutics. Anxiety symptoms is related to sensory hyperresponsiveness, and emerging evidence has shown that sensory atypicality in ASD could be contributed by the altered gut microbiota. Thus, intervention that targets the gut microbiota may improve the clinical anxiety symptoms in ASD children.

In this study, a pilot open-label trial will be conducted. It is planned that 30 ASD children who are below 12 years of age will be recruited from a regional children psychiatric specialist clinic to undergo a 12-week course of synbiotic. Feasibility, tolerability and preliminary efficacy of the synbiotic will be investigated using standardised parent-filled questionnaires. Changes in fecal microbiome and metabolites will be observed. The outcomes will be measured at weeks 6 and 12 of the 12-week course of synbiotic.

The results of the proposed study will provide insights with regards to the design and implementation of the main randomised controlled trial (RCT), contributing to the generation of evidence to the real-life efficacy the synbiotic. Physiological measurements of gut metagenomics and metabolomics will shed light on the specific mechanisms underlying clinical efficacies, which could inform the development of novel therapeutics targeting the microbiota-gut-brain axis in ASD.

ELIGIBILITY:
Inclusion Criteria:

1. ASD children of Chinese ethnicity aged <12 with diagnosis made by child psychiatrists based on Diagnostic and Statistical Manual, Fifth Edition (DSM-5) diagnostic criteria.
2. Elevated anxiety level, as measured by Anxiety Scale for Children-Autism Spectrum Disorder (ASC-ASD)
3. Presence of sensory hyperresponsiveness, as measured by Sensory Experience Questionnaire (SEQ)

Exclusion Criteria:

1. Co-occurring mental retardation, neurological, psychosis, depression or other severe mental illness.
2. History of non-functional gastrointestinal disorders such as inflammatory bowel disease and Hirschsprung's disease.
3. Presence of other significant physical illness, including but not limited to: current active malignancy, immunosuppression, organ failure and epilepsy
4. Exposure to antibiotics within 1 months of the study or history of using probiotics.
5. On special diet such as being a vegetarian

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and side effect | At week 6 and week 12 of the 12-week course of synbiotic
  Side effect, adverse events related to the 12-week course of synbiotic treatment

SECONDARY OUTCOMES:
Anxiety symptoms | At week 6 and week 12 of the 12-week course of synbiotic
  Change in anxiety symptoms during the12-week course of synbiotic treatment, as measured by the Anxiety Scale for Children-Autism Spectrum Disorder (ASC-ASD)
Sensory hyperresponsiveness | At week 6 and week 12 of the 12-week course of synbiotic
  Change in sensory hyperresponsiveness during the12-week course of synbiotic treatment, as measured by the Sensory Experience Questionnaire (SEQ)
Gastrointestinal symptoms | At week 6 and week 12 of the 12-week course of synbiotic
  Change in gastrointestinal symptoms during the12-week course of synbiotic treatment, as measured by the questionnaire on Paediatric Gastrointestinal Symptoms - Rome IV (QPGS-RIV).
Intestinal microbiota profile | At week 6 and week 12 of the 12-week course of synbiotic
  Stool samples will be collected for shotgun metagenomics sequencing to characterize the gut microbiota changes during the 12-week course of synbiotic treatment. Sequencing libraries will be prepared from extracted DNA and sequenced on an Illumina NovaSeq 6000 System. An average of 26 ± 3.3 million reads (6G data) per sample will be obtained 32 ± 4.6 million reads. Profiling of bacterial taxonomy and functional composition will be done with bioinformatic analysis Alpha-diversity indices, relative abundance of bacterial species will be quantified and compare across different timepoints of the study.
Intestinal metabolites profile | At week 6 and week 12 of the 12-week course of synbiotic
  Stool samples will be collected for metabolomics studies to characterize the gut metabolites changes during the 12-week course of synbiotic treatment. . In brief, the stool sample extracts were then separated using the Ultra Performance Liquid Chromatography. Skyline (MacLean et al., 2010) was used for metabolite identification and quantification. Following data normalization by probabilistic quotient normalization, principal component analysis on quality control samples that were analysed. Quantity of short-chained fatty acids, and other relevant metabolites will then be quantified and compare across different timepoints of the study

CONTACTS AND LOCATIONS:
Overall Officials: Wing Ho Wong, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No